CLINICAL TRIAL: NCT03074617
Title: Electromagnetic Field Effects of Mobile Communication (LTE) on Sleep in the Context of Genetic Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LTE-Sleep
Record Dates: First submitted 2017-02-23; First posted 2017-03-09 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTE field (Experimental)
  Interventions: Other: LTE field
- sham field (Sham Comparator)
  Interventions: Other: sham field

INTERVENTIONS:
Other: LTE field — electromagnetic field of the latest standard in mobile communication (long term evolution, LTE)
  Arms: LTE field
Other: sham field — no electromagnetic field
  Arms: sham field

SUMMARY:
The effect of electromagnetic fields of the latest standard in mobile communication (long term evolution, LTE) on sleep is studied in healthy, young individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* German knowledge (reading and writing)
* Right-handedness
* Body mass index (BMI) 18.5-25.0 kg/m2
* Mobile communication (phone calls) less than 2 hours per week
* Moderate alcohol consumption (less than 5 alcoholic beverages per week)
* Moderate caffeine consumption (less than 5 caffeinated foods per day, e.g. coke, coffee, energy drinks, green or black tea, chocolate)
* Informed consent

Exclusion Criteria:

* Travels across more than 2 time zones in the last 30 days or during the study
* Nocturnal shift work
* Extreme chronotype or extreme sleep duration (less than 5 hours or more than 10 hours on average)
* Sleep disorders or problems
* Severe acute or chronic neurological, mental or general health disorders, which might impair the participant's safety or affect the study's outcome
* Use of medication (regular or during the study), which might affect the study's outcome
* Recreational drug use
* Smoking (or other tobacco products)
* Severe skin allergies
* Relevant findings in physical examination or during the screening night (e.g. sleep disorders)
* Participation in an other clinical trial in the last 30 days or during the study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
electroencephalographic power during sleep after LTE exposure | up to 9 hours (approximately 11 p.m. to 8 a.m.)
  electroencephalogram (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Landolt, Principal Investigator — University of Zurich, Institute of Pharmacology and Toxicology
Locations (1):
- University of Zurich, Institute of Pharmacology and Toxicology, Zurich, Switzerland

REFERENCES:
- [Derived] Eicher C, Marty B, Achermann P, Huber R, Landolt HP. Reduced subjective sleep quality in people rating themselves as electro-hypersensitive: An observational study. Sleep Med. 2024 Jan;113:165-171. doi: 10.1016/j.sleep.2023.11.029. Epub 2023 Nov 21. PMID 38029625